CLINICAL TRIAL: NCT06651398
Title: To Dine or Not to Dine: Effect of Day-before Light Dinner on Bowel Cleansing Prior to Colonoscopy
Brief Title: A Study to Investigate the Effect of a Meal At 6pm the Day Before the Colonoscopy on the Bowel Cleansing with Plenvu
Acronym: DinNER1006
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Norgine BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S66191
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Bowel Preparation; Bowel Preparation for Colonoscopy; Bowel Cleansing for Colonoscopy; Healthy
Keywords: bowel preparation; colonoscopy preparation; bowel cleansing

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The endoscopist who performs the colonoscopy and the investigator who acts as second observer are blinded to objectively assess the BBPS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lenient diet (Experimental): This group can have a less stringent diet compared to the current standard of care and eat a light meal until 18h before drinking the first dose of the bowel preparation on the day before the colonoscopy
  Interventions: Behavioral: Lenient diet
- Control group (No Intervention): This group follows the strict diet similar to what is currently used in standard of care.

INTERVENTIONS:
Behavioral: Lenient diet — The interventional goup receives the lenient diet instructions and will eat a light meal until 18h on the day before the colonoscopy. The first dose of Plenvu will be started at 20h. All the other bowel preparation instructions will be the same as in the control group.
  Arms: Lenient diet

SUMMARY:
Bowel cleansing prior to colonoscopy is crucial to be able to perform a high-quality examination. Therefore maximum efforts are made to achieve optimal bowel cleansing including diet restriction and refraining from day-before dinner. However, the effect of this interdiction is currently not clear. On the other hand, patient compliance and experience with the entire procedure is important, especially for follow-up colonoscopies. Strict diets may interfere with this as an additional burden on the patient. In this study we want to assess whether a more lenient diet influences the quality of bowel preparation and whether it improves patient's experience.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for diagnostic colonoscopy
* Age between 40 and 85 years old
* Ability of normal oral ingestion
* Able to give informed consent by the patient or the legal representative

Exclusion Criteria:

* Participant has a history of (partial) colectomy, excluding appendectomy
* Inability of oral ingestion
* Chronic severe constipation, defined as the need for daily laxative use of any kind or the need to use laxatives to obtain defaecation.
* Uncontrolled coagulopathy
* Pregnancy
* Premenopausal women not adhering to any contraceptive method
* Inflammatory bowel disease
* Lynch syndrome
* Familial adenomatosis polyposis syndrome
* Serrated polyposis syndrome
* hypersensitivity to the active substances of PLENVU as listed in the SmPC section 6.1
* gastrointestinal obstruction or perforation
* ileus
* gastric emptying disorders (e.g. gastroparesis, gastric retention, etc.)
* phenylketonuria (due to the presence of aspartame in PLENVU)
* glucose-6-phosphate dehydrogenase deficiency (due to the presence of ascorbate in PLENVU)
* toxic megacolon
* Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an adequate bowel preparation (BBPS ≥6, and no segmental subscore ≤1) | Max 12 weeks

SECONDARY OUTCOMES:
Number of patients with an optimal bowel preparation (BBPS 8-9) | Max 12 weeks
Detection rates | Max 12 weeks
  Adenoma Detection Rate (ADR), Polyp Detection Rate (PDR), Serrated Polyp Detection Rate (SPDR), Advanced Adenoma Detection Rate (aADR)
Number of patients with high-quality right sided colon preparation (subscore = 3) | Max 12 weeks
Overall patient's tolerance, adherence and satisfaction based on the patient's diary | Max 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium